CLINICAL TRIAL: NCT03484234
Title: A Multi-center, Randomized, Study to Compare the Effectiveness of Sirolimus-eluting Stent (Ultimaster Stent) or Everolimus-eluting Stent (XIience Alpine Stent) for Long Coronary Lesions.
Brief Title: Percutaneous Treatment of LONG Native Coronary Lesions With Drug-Eluting Stent-VII: Sirolimus-eluting (Ultimaster) vs. Everolimus-Eluting Stents (Xience)
Acronym: LONG-DES VII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At sponsor's discretion : The purpose of study is no longer maintained
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2018-05
Record Dates: First submitted 2018-03-22; First posted 2018-03-30 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
Keywords: Drug eluting stent; everolimus eluting stent; sirolimus eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultimaster stent (Experimental)
  Interventions: Device: Ultimaster stent
- Xience alpine stent (Active Comparator)
  Interventions: Device: Xience alpine stent

INTERVENTIONS:
Device: Ultimaster stent — Percutaneous coronary intervention with Ultimaster stent for long lesion
  Arms: Ultimaster stent
Device: Xience alpine stent — Percutaneous coronary intervention with Xience alpine stent for long lesion
  Arms: Xience alpine stent

SUMMARY:
This study compares angiographic and clinical outcomes in patients with long coronary lesions treated with sirolimus-eluting stent (Ultimaster stent) or everolimus-eluting stent (Xience Alpine stent). The study uses a randomized, multicenter, controlled design approach.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 19 years of age.
2. Significant native coronary artery stenosis (>50% by visual estimate) with lesion length of more than 25mm, which requiring at long stent placement without intervening normal segment.
3. Patients with silent ischemia, stable or unstable angina pectoris, ad Non-ST-elevation myocardial infarction (NSTEMI)
4. The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Any contraindication to any of the following medications: aspirin, heparin, clopidogrel, stainless steel, contrast agents, sirolimus, or everolimus
2. An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 6 months post enrollment.
3. Acute ST-segment-elevation MI or cardiogenic shock
4. Terminal illness with life expectancy <1 year
5. In-stent restenosis at target vessel (either bare metal stent or drug-eluting stent segment). However, non-target vessel ISR is permitted.
6. Patients with EF<30%.
7. Serum creatinine level ≥ 2.0mg/dL or dependence on dialysis.
8. Patients with left main stem stenosis (>50% by visual estimate)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
In-segment late luminal loss | 13-month

SECONDARY OUTCOMES:
All death | 1 year
Cardiac death | 1 year
Myocardial infarction (MI) | 1 year
Composite of death or MI | 1 year
Composite of cardiac death or MI | 1 year
Target vessel revascularization (ischemia-driven and clinically-driven) | 1 year
Target lesion revascularization (ischemia-driven and clinically-driven) | 1 year
Target-vessel failure | 1 year
  death from any cause, myocardial infarction, and ischemic-driven target-vessel revascularization
Stent thrombosis | 1 year
In-stent late loss | 13-month
  In-stent late loss at 13-month angiographic follow-up
In-stent and in-segment restenosis | 13-month
  In-stent and in-segment restenosis at 13-month angiographic follow-up
Angiographic pattern of restenosis | 13-month
  Angiographic pattern of restenosis at 13 -month angiographic follow-up
Volume of intimal hyperplasia | 13-month
  Volume of intimal hyperplasia at 13-month IVUS follow-up (sub-study)
Incidence of late stent malapposition | 13-month
  Incidence of late stent malapposition at 13-month IVUS follow-up (sub-study)
Procedural success | 5 days
  Procedural success defined as achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or repeat revascularization of the target lesion during the hospital stay.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Gangwon National Univ. Hospital, Chuncheon
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided